CLINICAL TRIAL: NCT06393686
Title: Impact of Yoga Intervention on Physical Fitness Parameters in Preadolescent Children: A Randomized Controlled Trial
Brief Title: The Effect of Yoga on the Fitness of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Melis Bagkur, assist prof, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YDU/2019/74-938
Record Dates: First submitted 2024-04-17; First posted 2024-05-01 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Exercise Test; Physical Endurance; Muscles
Keywords: Yoga; Muscle Stretching Exercises; Physical Endurance
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CONTROLLED TRIAL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): The yoga intervention will be implemented every two weeks, with each session lasting 45 minutes and implemented for 10 weeks. Sessions will always be led by the same certified yoga instructor. Each session will include a variety of different yoga poses, as well as breathing techniques and deep relaxation methods.
  Interventions: Other: yoga
- Control Group (No Intervention): There will be no intervention in the control group.

INTERVENTIONS:
Other: yoga — The yoga intervention will be implemented every two weeks, with each session lasting 45 minutes and implemented for 10 weeks. Sessions will always be led by the same certified yoga instructor. Each session will include a variety of different yoga poses, as well as breathing techniques and deep relaxation methods.
  Arms: Yoga Group

SUMMARY:
This study aims to evaluate the effect of yoga on physical fitness among healthy primary school children using a randomized control design. A total of 52 children, ages 8-13, will be randomly assigned to either the Yoga Group or the Control Group. Participants will be assessed using the EUROFIT Test Battery as the primary outcome measure.

The Yoga Group will do 45-minute yoga sessions twice a week for 10 weeks, while the Control Group will not receive any intervention. Outcome assessments will be repeated at the end of the 10-week intervention period.

DETAILED DESCRIPTION:
This investigation is a randomized controlled trial designed to assess the physical fitness levels among primary school-age children subjected to diverse yoga interventions, comparing them with the outcomes observed in a control group devoid of such interventions.The study encompasses a 10-week intervention phase, during which participants undergo evaluation at two specific time points: Initial assessment (M1), conducted one week preceding the commencement of the exercise program, and subsequent evaluation (M2), executed one week post the conclusion of the program.Anthropometric measurements will determine the height of the participants using a non-elastic measuring tape (SECA brand) attached to the wall. Body Mass Index (BMI) will be calculated with the Tanita MC-180MA III device.The physical fitness of children will be measured with the Eurofit test battery.

ELIGIBILITY:
Inclusion Criteria:

* Participants who do not have any mental or physical disabilities
* Participants who have not participated in any exercise regime for the previous six months

Exclusion Criteria:

• Individuals who do not participate in 90 percent of the 10-week yoga training program.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
EUROFIT Test Battery | 12 weeks
  The 10 tests for the Eurofit Test Battery are used as standards in the measurements of school-aged children.
  Anthropometry: Height, Weight, BMI, Skinfold thickness
  * Flamingo balance test
  * Arm movement speed
  * Sit and reach
  * Standing long jump
  * Hand grip strength
  * 30s Shuttle Bent arm hanging
  * 10 x 5 meter shuttle run
  * 20 m endurance (shuttle) run
Anthropometric measurements | 12 weeks
  Anthropometric measurements involved determining participants' height using a non-elastic measuring tape (SECA brand), affixed to a wall. The Tanita MC-180MA III device facilitated weight analysis, and Body Mass Index (BMI) (kg/m2) was calculated by dividing body weight (in kilograms) by the square of height (in meters).
Body Mass Index | 12 weeks
  Weight in kilograms and height in meters will been calculated and, weight and height will be combined to report BMI in kg/m2.

CONTACTS AND LOCATIONS:
Locations (1):
- Near East University, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No